CLINICAL TRIAL: NCT01147393
Title: Phase I/II Study of Combination Veltuzumab (Anti-CD20) and Fractionated 90Y- Epratuzumab (Anti-CD22) Radioimmunotherapy in Patients With Follicular Lymphoma
Brief Title: Combination Veltuzumab and Fractionated 90Y- Epratuzumab Radioimmunotherapy in Follicular Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: closed to enrollment due to slow patient accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1001010838
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — veltuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): two weekly infusions of 90Y-epratuzumab tetraxetan in combination with four weekly infusions of 200 mg/m2 veltuzumab.
  Interventions: Drug: 90Y-epratuzumab tetraxetan; Biological: veltuzumab

INTERVENTIONS:
Drug: 90Y-epratuzumab tetraxetan — The 90Y-epratuzumab treatment will begin one week after the 4th veltuzumab injection. Patients will receive unlabeled, unconjugated epratuzumab (1.5 mg/kg) that will be infused over ~30 minutes. All patients will then receive a 90Y-epratuzumab dose. Dose will be escalated by patient cohort either at 15 mCi/m2 or 20 mCi/m2. The second 90Y-epratuzumab treatment will be given at the same dose, 1 week after the first 90Y-epratuzumab dose.
Biological: veltuzumab — Veltuzumab is given in 4 weekly doses, each 200 mg/m2.

SUMMARY:
A Phase I/II clinical trial using a fractionated dosing regimen of 90Y-epratuzumab (anti-CD22) has showed encouraging responses in follicular and aggressive NHL with an ability to administer safely 2 injections of 20 mCi/m2 spaced 1 week apart. The investigators propose to combine this active 90Y-epratuzumab treatment with a regimen of veltuzumab that was also found active in Phase I/II trials.

The goal of this study is to determine the safety and efficacy of 90Y-epratuzumab when used in combination with veltuzumab. The primary objective is to determine the response rate of this combination treatment. Secondary objectives are to assess safety, pharmacokinetics and targeting of 90Y-epratuzumab . Veltuzumab blood levels and anti-antibody responses will also be monitored at various times.

DETAILED DESCRIPTION:
The treatment regimen consists of 2 elements. The first element is represented by one courses of veltuzumab (4 weekly injections of 200 mg/m2). 90Y-epratuzumab will be given as 2 injections at escalating doses 1 week apart and administered starting one week following the 4th veltuzumab injection.

After confirming eligibility and undergoing baseline assessments, the treatment starts with an imaging study using 111In-epratuzumab (5-mCi 111In-DOTA-epratuzumab co-infused with a total of 1.5 mg/kg unlabeled epratuzumab). Blood samples (~7 samples, 5 mL each) for pharmacokinetic analysis will be collected over 5-7 days, and patients will be imaged on 4 separate occasions (e.g., the day of injection (Day 0), Day 1, Day 3, 4, or 5, and day 6 or 7).

The patient will then initiate veltuzumab treatments starting 7 days after the 111In-epratuzumab injection. Veltuzumab is given in 4 weekly doses, each 200 mg/m2. A single blood sample will be taken before each veltuzumab dose to assess residual veltuzumab concentrations in the serum, and then at 1 h later to determine peak values. Patients will receive unlabeled, unconjugated epratuzumab (1.5 mg/kg) that will be infused over ~30 minutes. Patients will also receive 111In-epratuzumab immediately following the unlabeled epratuzumab. Blood samples will be collected at the same intervals as after the first 111In-epratuzumab. Only 2 imaging sessions will be required, on Day 1 and then again on day 6 or 7 (these days should match those obtained after the first 111In-epratuzumab injection).

The 90Y-epratuzumab treatment will begin one week after the 4th veltuzumab injection. Patients will receive unlabeled, unconjugated epratuzumab (1.5 mg/kg) that will be infused over ~30 minutes. All patients will then receive a 90Y-epratuzumab dose. Dose will be escalated by patient cohort starting at 2x15 mCi/m2 and, at 2x 20 mCi/m2, and 2x 25 mCi/m2.. Blood samples will be collected at the same intervals as after each 111In-epratuzumab.Patients will also receive 111In-epratuzumab immediately following the unlabeled epratuzumab and immediately before the 90Y-epratuzumab injection. Blood samples will be collected at the same intervals as after the first 111In-epratuzumab. Only 2 imaging sessions will be required, on Day 1 and then again on day 6 or 7 (these days should match those obtained after the first 111In-epratuzumab injection).

The second 90Y-epratuzumab treatment will be given at the same dose, 1 week after the first 90Y-epratuzumab dose. CBC will be checked prior to administration of this second dose to ensure blood counts continue to meet criteria for treatment as specified in inclusion criteria. Blood samples will again be collected over the same period as the first injection, but no imaging studies are required.

Patients are closely monitored during all infusions, and then at intervals over a 12-weeks post-treatment evaluation period, with evaluation procedures including vital signs, physical examination, CT (chest, abdomen, pelvis, other regions of involvement), CBC, serum chemistries, serum immunoglobulins, urinalysis, peripheral blood B-cell levels (immunophenotyping based on CD19), and serum samples for HAHA (veltuzumab and epratuzumab ELISA to be analyzed by Immunomedics). Follow-up evaluations then continue every 3 months for up to 5 years or until progression occurs or until resolution of treatment-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years old
* Histological diagnosis of CD20+ Follicular lymphoma by WHO lymphoma criteria.
* FLIPI intermediate or high risk (2-5 risk factors)
* No prior systemic treatment for NHL
* Measurable disease by CT, with at least one lesion >1.5 cm in one dimension
* Life expectancy of at least 6 months
* ECOG performance status > = 2
* Patients must have normal organ and marrow function as defined below:

  * ANC > = 1,500/uL
  * platelets > = 100,000/uL
  * total bilirubin < = 1.5 x upper limit of normal
  * AST(SGOT)/ALT(SGPT) < = 2.5 X upper limit of normal
  * creatinine < = 1.5 x upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study until at least 12 weeks after the last weekly veltuzumab infusion.
* Primary CNS lymphoma, HIV lymphoma or transformed lymphoma, or presence of symptomatic CNS metastases or carcinomatous meningitis.
* Bulky disease by CT, defined as any single mass >10 cm in its greatest diameter
* Disease status eligible for potentially curative external beam radiation (stage 1 or contiguous stage 2 at sites appropriate for radiotherapy)
* Bone marrow involvement ≥25%; patients with CLL
* Pleural effusion with positive cytology for lymphoma
* Patients known to be HIV positive or hepatitis B positive
* Corticosteroid use within 2 weeks, unless 20 mg/day or less at stable dose.
* Prior malignancy with less than a 1-year disease-free interval, excluding non-melanoma skin cancers and carcinoma in situ of the cervix.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-08-06 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Dose Level 1
Arm/Group | All Subjects
Started | 3
Completed | 1
Not Completed | 2
Not completed — Dose limiting Toxicity | 2
Period: Dose Level -1
Arm/Group | All Subjects
Started | 1
Completed | 0
Not Completed | 1
Not completed — Dose Limited Toxicity | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  Patients by Age: 60-69 Years of Age | 3
  Patients by Age: 70-79 Years of Age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine the Maximum Tolerated 90Y Dose
Population: Data was not collected
Arm/Group | All Subjects
Number analyzed (Participants) | 0

2. Primary Outcome: Dose-limiting Toxicity
Description: NCI CTC version 3.0 is used to grade all adverse events and to provide management guidelines for infusional toxicity. Dose-limiting toxicity (DLT) is defined as follows:
  Hematologic: Grade 4 toxicity >7 days, as specified by hemoglobin levels, platelet counts or absolute neutrophil count (ANC) or failure of hemoglobin levels, platelet counts or ANC to recover to Grade 1 levels within 12 weeks of completing the treatment cycle (with the use of RBC and platelet transfusions or growth factors during the 12 weeks if necessary, but at least one week without any support prior to qualifying Grade 1 levels).
  Non-Hematologic: Any Grade 3 or Grade 4. Other: Any Grade 2 autoimmune reactions, or the occurrence of Grade 2 immediate-type allergic/hypersensitivity reactions (e.g., urticaria, wheezing, hypoxia and dyspnea) will be considered DLT and will also require the infusion to be permanently terminated.
  Occurrence of DLT requires a patient's treatment to be permanently discontinued
Population: Data were not collected
Arm/Group | All Subjects
Number analyzed (Participants) | 0

3. Primary Outcome: Safety
Population: Data was not evaluated
Arm/Group | All Subjects
Number analyzed (Participants) | 0

4. Primary Outcome: The Primary Objective of the Phase II Portion of the Study is to Determine the Anti-tumor Efficacy, as Measured by Response Rate, of Fractionated 90Y-epratutumab IgG Given in Combination With Veltuzumab Anti-CD20 IgG Therapy
Population: Data were not collected
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Dose Level 1: veltzumab: 200 mg/m2 Unconjugated epratuzumab: 1.5 mg/kg 111-In-epratuzumab: 5 mCi 90-Y-epratuzumab: 15 mCi/m2
- Dose Level -1: veltzumab: 200 mg/m2 Unconjugated epratuzumab: 1.5 mg/kg 111-In-epratuzumab: 5 mCi 90-Y-epratuzumab: 10 mCi/m2
Arm/Group | Dose Level 1 | Dose Level -1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level -1 (N=1)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 1 (3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (6) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hives (infusion reaction) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Flutters (neck and throat) (General disorders) | 1 (1) | 0 (0)
Taste alteration (General disorders) | 1 (1) | 0 (0)
Easy bruisability (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding gums (General disorders) | 1 (1) | 0 (0)
Nasal congestion (General disorders) | 1 (1) | 0 (0)
Cough (General disorders) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Dyspnea (General disorders) | 2 (3) | 1 (1)
Insomnia (General disorders) | 3 (4) | 0 (0)
Nausea (General disorders) | 2 (2) | 1 (1)
Sore throat (General disorders) | 2 (2) | 0 (0)
Flatulence (General disorders) | 2 (2) | 0 (0)
Hyperpigmentation (tongue) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Visual changes (aura) (General disorders) | 1 (1) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain (groin) (General disorders) | 1 (1) | 0 (0)
Cyst (outer labia) (General disorders) | 1 (1) | 0 (0)
Pruritic rash (left shoulder,chest) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 0 (0)
Pain (left unla, radial head fracture) (General disorders) | 1 (1) | 0 (0)
Ear congestion (General disorders) | 1 (1) | 0 (0)
Heartburn (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Diplopia (General disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Pain (joint) (General disorders) | 1 (1) | 0 (0)
Neuropathy (numbness, tingling) (Nervous system disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Heat intolerance (General disorders) | 1 (1) | 0 (0)
Cold intolerance (General disorders) | 1 (1) | 0 (0)
Joint function (stiffness) (General disorders) | 1 (1) | 0 (0)
Orthopnea (General disorders) | 1 (1) | 0 (0)
Hyperpigmentation (hands, fingers) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (leg) (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Constipation (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes